CLINICAL TRIAL: NCT07163208
Title: Therapeutic Efficacy of Different Wavelengths of Low-Level Laser Therapy in the Treatment of Cervicogenic Headache
Acronym: WELL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Arooj Munawar, Principal Investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 520/24
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic Headache; Low-Level Laser Therapy; Neck Pain
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Three parallel groups receive different LLLT wavelengths (675nm, 820nm, 46-cluster LED) plus routine physical therapy, assessed at baseline, 3 weeks, 6 weeks, and follow-ups
Who Masked: Participant, Outcomes Assessor
Masking Description: In addition to participants and outcomes assessors being masked, care providers administering the low-level laser therapy (LLLT) interventions are also blinded to the specific wavelength or modality (675nm, 820nm, or 46-cluster LED probe) assigned to each group to minimize bias in treatment delivery, ensuring the study's integrity across all three parallel experimental groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: 675nm LLLT + RPT (Experimental): Single direct in-contact pencil probe, wavelength 675 nm, power 30 mW. Irradiance 222 mW/cm², fluence 6.7 J/cm², spot size 0.9 cm². Delivered in continuous and pulsed (2.5 Hz) modes, 6 Joules for 30 sec per treatment point (lymphatic chain, sub-occipital musculature, facet joints, nerve root exits, trigger points). Administered 3× weekly for 6 weeks (30 min/session).
  Device: Omega XP Model, Omega Laser Systems (UK) Class II therapeutic photobiomodulation device. Equipped with single direct in-contact pencil probes (675 nm, 30 mW; 820 nm, 200 mW) and a 46-cluster LED probe (mixed diodes 660-950 nm). Operates in continuous and pulsed (2.5 Hz) modes. Spot size 0.9-10 cm², irradiance 95-222 mW/cm², fluence 6.7-11.4 J/cm². CE-certified for therapeutic use; applied in this trial for cervicogenic headache management.
  Interventions: Device: Low-Level Laser Therapy (LLLT); Other: Routine Physical Therapy (RPT)
- Group 2: 820nm LLLT + RPT (Experimental): Single direct in-contact pencil probe, wavelength 820 nm, power 200 mW. Irradiance 222 mW/cm², fluence 6.7 J/cm², spot size 0.9 cm². Delivered in continuous and pulsed (2.5 Hz) modes, 6 Joules for 30 sec per treatment point (same anatomical sites as Group 1). Administered 3× weekly for 6 weeks (30 min/session).
  Device: Omega XP Model, Omega Laser Systems (UK) Class II therapeutic photobiomodulation device. Equipped with single direct in-contact pencil probes (675 nm, 30 mW; 820 nm, 200 mW) and a 46-cluster LED probe (mixed diodes 660-950 nm). Operates in continuous and pulsed (2.5 Hz) modes. Spot size 0.9-10 cm², irradiance 95-222 mW/cm², fluence 6.7-11.4 J/cm². CE-certified for therapeutic use; applied in this trial for cervicogenic headache management.
  Interventions: Device: Low-Level Laser Therapy (LLLT); Other: Routine Physical Therapy (RPT)
- Group 3: 46 Cluster LED Probe + RPT (Experimental): 46-cluster LED probe combining 660 nm, 950 nm, 870 nm, 880 nm, 940 nm, 820 nm. Irradiance 95 mW/cm², fluence 11.4 J/cm², spot size 10 cm². Delivered in continuous and pulsed (2.5 Hz) modes, 114 Joules for 120 sec per treatment area (same anatomical sites as above). Administered 3× weekly for 6 weeks (30 min/session).
  Device: Omega XP Model, Omega Laser Systems (UK) Class II therapeutic photobiomodulation device. Equipped with single direct in-contact pencil probes (675 nm, 30 mW; 820 nm, 200 mW) and a 46-cluster LED probe (mixed diodes 660-950 nm). Operates in continuous and pulsed (2.5 Hz) modes. Spot size 0.9-10 cm², irradiance 95-222 mW/cm², fluence 6.7-11.4 J/cm². CE-certified for therapeutic use; applied in this trial for cervicogenic headache management.
  Interventions: Device: Low-Level Laser Therapy (LLLT); Other: Routine Physical Therapy (RPT)

INTERVENTIONS:
Device: Low-Level Laser Therapy (LLLT) — Low-level laser therapy using the Omega XP Model with wavelengths of 675nm (30mW), 820nm (200mW), or 46-cluster LED probe (mixed wavelengths: 660nm, 950nm, 870nm, 880nm, 940nm, 820nm), applied three times weekly for 30 minutes over 6 weeks to target cervical lymphatic chain, musculature, and trigger points for pain relief in cervicogenic headache.
Other: Routine Physical Therapy (RPT) — Warm-up: Active cervical ROM (5-10 reps, pain-free range). Stretching: Upper trapezius, levator scapulae, SCM; hold 15-30 sec, 3-5 reps, NRS ≤ 3/10. Therapeutic exercises: cervical deep flexors, scapular stabilization (2-3 sets × 10-15 reps, Borg 11-13), progressed weekly. Modalities: Hot pack 15 min at 40-45°C; TENS 80-100 Hz, 50-100 µs pulse width, 20 min. Frequency: 3× weekly for 6 weeks. Safety: contraindications screened; pain/exertion monitored pre/post.

SUMMARY:
This study tests if low-level laser therapy (LLLT) with different light wavelengths can help people with cervicogenic headache, a type of headache caused by neck problems. Adults aged 18-65 with this headache for at least 3 months will try one of three LLLT treatments (675nm, 820nm, or a mix of wavelengths) along with regular physical therapy like stretching and exercises. The study will check pain levels, how often headaches happen, neck movement, disability, and quality of life over 6 weeks, with follow-ups at 3 and 6 months. the investigators want to find the best LLLT option to reduce headache symptoms safely.

DETAILED DESCRIPTION:
This single-center, single-blinded randomized clinical trial investigates the therapeutic efficacy of low-level laser therapy (LLLT) at different wavelengths-675nm (30mW), 820nm (200mW), and a 46-cluster LED probe (combining 660nm, 950nm, 870nm, 880nm, 940nm, 820nm)-in treating cervicogenic headache (CGH), a secondary headache originating from cervical spine dysfunction. Conducted at the Department of Physiotherapy, Sir Ganga Ram Hospital, Lahore, the study spans 18 months post-BASR approval, with a 6-week intervention period and 6-month follow-up. Participants are randomized into three parallel groups, each receiving LLLT (using the Omega XP Model) plus routine physical therapy (stretching, exercise, hot pack, TENS) three times weekly for 30 minutes over 18 sessions. The trial aims to compare the effectiveness of these modalities in reducing pain (VAS), headache frequency (diary), cervical range of motion (goniometry), neck disability (NDI), quality of life (SF-36), and forward head posture (camera). Ethical approval was granted by The University of Lahore's Research Ethical Committee (Ref: REC-UOL-/520/08/24, dated 05-09-2024), ensuring participant consent and confidentiality. The study addresses a research gap in wavelength-specific LLLT efficacy for CGH, potentially guiding future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years diagnosed with cervicogenic headache based on the International Classification of Headache Disorders (ICHD-3) criteria.
* Persistent headaches for at least 3 months.
* No previous exposure to low-level laser therapy (LLLT).

Exclusion Criteria:

* Patients with other primary headache disorders (e.g., migraine, tension-type headache).
* History of cervical spine surgery.
* Pregnant or lactating women.
* Patients with a history of photosensitivity or taking photosensitizing medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Reduction in Headache Frequency | Baseline, 3 weeks, 6 weeks, 3 months, 6 months
  Measured by patient diary recording
Mean Change in Pain Intensity (VAS Score, 0-10) | Baseline, 3 weeks, 6 weeks, 3 months, 6 months
  Measured by Visual Analog Scale (VAS, 0-10)

SECONDARY OUTCOMES:
Change in Cervical ROM (degrees) | Baseline, 3 weeks, 6 weeks, 3 months, 6 months
  Measured by universal goniometer
Mean Difference in Neck Disability Index (NDI) Score | Baseline, 3 weeks, 6 weeks, 3 months, 6 months
  Measured by Neck Disability Index (NDI, Urdu version)
Mean Change in SF-36 Quality of Life Score | Baseline, 3 weeks, 6 weeks, 3 months, 6 months
  Measured by Short Form Health Survey (SF-36)
Change in Forward Head Posture (degrees, camera-based measurement) | Baseline, 3 weeks, 6 weeks, 3 months, 6 months
  Measured by mobile camera picture, degree

CONTACTS AND LOCATIONS:
Overall Officials: Umair Ahmed, PhD, Study Director — University of Lahore, Lahore, Pakistan
Locations (1):
- Department of Physiotherapy, Sir Ganga Ram Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome results will be shared, including baseline demographic and clinical characteristics, pain scores (VAS), headache frequency, Neck Disability Index (NDI), cervical ROM, SF-36 quality of life measures, and forward head posture assessments.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will be available beginning 6 months after publication of the main trial results and will remain accessible for 5 years thereafter.
Access Criteria: Qualified researchers affiliated with academic institutions or healthcare organizations may request access. Proposals will be reviewed by the principal investigator and supervisory team to ensure scientific merit and compliance with ethical approvals. Data will be shared in de-identified format only through a secure data repository (encrypted file transfer or institutional repository) after signing a data-sharing agreement.

REFERENCES:
- [Background] Bjordal JM, Johnson MI, Iversen V, Aimbire F, Lopes-Martins RA. Low-level laser therapy in acute pain: a systematic review of possible mechanisms of action and clinical effects in randomized placebo-controlled trials. Photomed Laser Surg. 2006 Apr;24(2):158-68. doi: 10.1089/pho.2006.24.158. PMID 16706694